CLINICAL TRIAL: NCT02671539
Title: THOR - Tübingen Choroideremia Gene Therapy Trial Open Label Phase 2 Clinical Trial Using an Adeno-associated Viral Vector (AAV2) Encoding Rab-escort Protein 1 (REP1)
Brief Title: THOR - Tübingen Choroideremia Gene Therapy Trial
Acronym: THOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: STZ eyetrial (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THOR-TUE-01
Record Dates: First submitted 2016-01-19; First posted 2016-02-02 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Choroideremia
Keywords: gene therapy; hereditary retinal degeneration; rAAV2.REP1
MeSH Terms: conditions — Choroideremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open label injection of rAAV2.REP1 (Experimental): This is an open label, single arm interventional trial with subretinal injection of rAAV2.REP1 and fellow eye comparison
  Interventions: Genetic: rAAV2.REP1

INTERVENTIONS:
Genetic: rAAV2.REP1 — single subretinal injection

SUMMARY:
An open label monocentric phase II trial in adult males with a clinical phenotype of choroideremia and a confirmed molecular diagnosis of a null mutation in the gene encoding REP1 to assess the anatomical and functional outcomes, as well as the safety of a single subretinal injection of rAAV2.REP1 in 6 subjects with genetically confirmed choroideremia for up to 24 months.

DETAILED DESCRIPTION:
Study name: THOR - Tübingen Choroideremia gene therapy trial open label Phase 2 clinical trial using an adeno-associated viral vector (AAV2) encoding Rab-escort protein 1 (REP1)

Phase: Phase II

Indication: Adult males with a clinical phenotype of choroideremia and a confirmed molecular diagnosis of a null mutation in the gene encoding REP1

Aim of study: To assess the anatomical and functional outcomes, as well as the safety of a single subretinal injection of rAAV2.REP1 in subjects with genetically confirmed choroideremia for up to 24 months.

Primary Endpoint: Change from baseline in best corrected visual acuity in treated eye, compared to untreated control eye

Study design: Open label monocenter study

Study population: 6 male adults affected by choroideremia

Inclusion Criteria

1. Participant is willing and able to give informed consent for participation in the study.
2. Male aged 18 years or above.
3. Genetically confirmed diagnosis of choroideremia. Patients without a confirmed mutation in the CHM gene, but who have the clinical phenotype typical of choroideremia can only be enrolled if they meet all the following three criteria: (i) family history consistent with X-linked inheritance, (ii) absent REP1 protein on Western blot of a blood sample and, (iii) normal RPE65 gene on sequencing.
4. Active disease visible clinically within the macula region
5. Best-corrected visual acuity equal to or worse than 6/9 (20/32; Decimal 0.63; LogMAR 0.2) but better than or equal to 6/60 (20/200; Decimal 0.1; LogMAR 1.0) in the study eye.

Exclusion Criteria

1. Female and child participants (under the age of 18)
2. Participants with a history of amblyopia in the study eye
3. Men unwilling to use barrier contraception methods, if relevant
4. Absence of quantifiable visual function in the fellow eye or other ocular morbidity which might confound use of the fellow eye as a long-term control.
5. Any other significant ocular and non-ocular disease/disorder or retinal surgery which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the results of the study, or the participant's ability to participate in the study. This would include not taking or having a contraindication to oral prednisolone, such as a history of gastric ulcer or significant side effects.
6. Participants who have participated in another research study involving an investigational product in the past 12 weeks, or having had gene or cellular therapy at any time prior to this study.
7. Patients with amblyopic eyes should be excluded in general, since the evaluation of the primary endpoint presupposes the ability to fixate both eyes
8. Prior intraocular surgery within six months
9. Intolerance to local anesthesia and/or contraindication to IVT surgery (anemia Hb<8g/dl, severe cardiovascular disease, severe coagulopathy, etc.)
10. High fever or high fever disease, patients with a history of autoimmune conditions/ other systemic diseases that may have ocular manifestations (e.g. sarcoidosis) or neurodegenerative conditions (e.g. multiple sclerosis, neuromyelitis optica, Parkinson's disease)
11. Patients suffering from other genetic mutations leading to pathological retinal conditions
12. Patients treated by oral corticoids within 14 days prior inclusion at the study entry

Patient number: 6

Treatment: Each participant will receive a single treatment of the rAAV2.REP1 vector (0.1ml containing 1011 AAV2 genome particles) administered by subretinal injection during a vitrectomy operation. No placebo will be used. ln order to minimize selection bias both eyes are randomized to either treatment or control.

Main criteria: Primary endpoint: Change from baseline in best corrected visual acuity in treated eye, compared to untreated control eye up to 24 months after vector administration Secondary endpoints: Absence of vector related adverse reactions 24 months after vector administration. Demonstration of improved retinal anatomy and/or visual function other than best corrected visual acuity in treated eye compared to the untreated control eye 24 months after vector administration.

Statistical methods:

Summary statistics will be presented for both eyes (Treated Eye versus Control Eye groups). No formal statistical comparison will be performed (no p-value will be computed). For categorical/binary data, the number and proportion of patients in each category will be presented with its 95% Confidence Interval (CI). For continuous data, mean (and its 95% CI) and Standard Deviation (SD) will be presented.

The primary outcome measure will be the proportion of patients with a relative change from baseline of > 5 in ETDRS letters (treated vs. untreated eye, change from BL). At each time point, the change from baseline in ETDRS letters will be computed for each eye. The mean change from baseline in ETDRS letters will be presented for both the treated eye and the control eye groups.

At each time point, the change from baseline and the percentage change from baseline in the area of autofluoresence will be computed for each eye and their mean will be presented for both the treated eye and the control eye groups.

With regards to microperimetry, at each time point, the change from baseline in mean sensitivity will be computed for each eye. The mean change from baseline in mean sensitivity will be presented for both the treated eye and the control eye groups.

Adverse events will be listed. Other Investigator Sponsored Studies are expected to be run with a similar protocol for the same indication and with the same intervention. A meta-analysis on the Investigator Sponsored studies is planned. A separate Statistical Analysis Plan describing the details of the meta-analysis will be developed.

Timetable:

Planned trial period: 24 month Follow-up duration: 36 month

The end of trial is the date on which the last treated patient completes the tests of their planned close-out visit.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent for participation in the study.
2. Male aged 18 years or above.
3. Genetically confirmed diagnosis of choroideremia. Patients without a confirmed mutation in the CHM gene, but who have the clinical phenotype typical of choroideremia can only be enrolled if they meet all the following three criteria: (i) family history consistent with X-linked inheritance, (ii) absent REP1 protein on Western blot of a blood sample and, (iii) normal RPE65 gene on sequencing.
4. Active disease visible clinically within the macula region
5. Best-corrected visual acuity equal to or worse than 6/9 (20/32; Decimal 0.63; LogMAR 0.2) but better than or equal to 6/60 (20/200; Decimal 0.1; LogMAR 1.0) in the study eye.

Exclusion Criteria:

1. Female and child participants (under the age of 18)
2. Participants with a history of amblyopia in the study eye
3. Men unwilling to use barrier contraception methods, if relevant
4. Absence of quantifiable visual function in the fellow eye or other ocular morbidity which might confound use of the fellow eye as a long-term control.
5. Any other significant ocular and non-ocular disease/disorder or retinal surgery which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the results of the study, or the participant's ability to participate in the study. This would include not taking or having a contraindication to oral prednisolone, such as a history of gastric ulcer or significant side effects.
6. Participants who have participated in another research study involving an investigational product in the past 12 weeks, or having had gene or cellular therapy at any time prior to this study.
7. Patients with amblyopic eyes should be excluded in general, since the evaluation of the primary endpoint presupposes the ability to fixate both eyes
8. Prior intraocular surgery within six months
9. Intolerance to local anesthesia and/or contraindication to IVT surgery (anemia Hb<8g/dl, severe cardiovascular disease, severe coagulopathy, etc.)
10. High fever or high fever disease, patients with a history of autoimmune conditions/ other systemic diseases that may have ocular manifestations (e.g. sarcoidosis) or neurodegenerative conditions (e.g. multiple sclerosis, neuromyelitis optica, Parkinson's disease)
11. Patients suffering from other genetic mutations leading to pathological retinal conditions
12. Patients treated by oral corticoids within 14 days prior inclusion at the study entry

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
best corrected visual acuity in treated eye | up to 24 months after vector administration
  Change from baseline in best corrected visual acuity in treated eye, compared to untreated control eye up to 24 months after vector administration

SECONDARY OUTCOMES:
Absence of vector-related adverse reactions | 24 months after vector administration
fundus autofluorescence analysis | 24 months after vector administration
  improved retinal anatomy in treated eye compared to the untreated control eye 24 months after vector administration
central visual field using microperimetry readings | 24 months after vector administration
  improved visual function in treated eye compared to the untreated control eye 24 months after vector administration
contrast sensitivity | 24 months after vector administration
  improved visual function other than best corrected visual acuity in treated eye compared to the untreated control eye 24 months after vector administration (scale)
colour vision | 24 months after vector administration
  improved visual function other than best corrected visual acuity in treated eye compared to the untreated control eye 24 months after vector administration (physiological parameter)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel D Fischer, MD, PhD, Principal Investigator — Centre for Ophthalmology, University Hospital Tübingen, Germany
Locations (1):
- University Hospital Tuebingen, Center for Ophthalmology, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fischer MD, Ochakovski GA, Beier B, Seitz IP, Vaheb Y, Kortuem C, Reichel FFL, Kuehlewein L, Kahle NA, Peters T, Girach A, Zrenner E, Ueffing M, MacLaren RE, Bartz-Schmidt KU, Wilhelm B. Efficacy and Safety of Retinal Gene Therapy Using Adeno-Associated Virus Vector for Patients With Choroideremia: A Randomized Clinical Trial. JAMA Ophthalmol. 2019 Nov 1;137(11):1247-1254. doi: 10.1001/jamaophthalmol.2019.3278. PMID 31465092